CLINICAL TRIAL: NCT06041958
Title: Effects of Extracorporeal Shock Wave Therapy and Pulse Electromagnetic Field Therapy on Lymphoedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zheng-Yu Hoe, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Zheng-Yu Hoe, MD., PhD., Principal Investigator, Kaohsiung Veterans General Hospital.
Organization: Kaohsiung Veterans General Hospital. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-CT12-01(210917-1)
Record Dates: First submitted 2023-08-31; First posted 2023-09-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Extracorporeal Shockwave Therapy; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- General rehabilitation therapy (Active Comparator): Conducting a general rehabilitation program for lymphedema, three times a week, continuing until the end of the experiment.
  Interventions: Other: Rehabilitation
- ESWT therapy group (Experimental): Participants are randomly assigned to receive either shockwave therapy or electromagnetic pulse therapy. Once assigned, the treatment method is fixed and continues for 12 weeks. From week 1 to week 12, participants receive either extracorporeal shockwave therapy or electromagnetic pulse therapy three times a week, totaling 36 sessions. After the completion of the 12-week treatment, the general rehabilitation program for lymphedema continues, conducted three times a week.
  Interventions: Device: Extracorporeal shock wave therapy
- PEMFT therapy group (Experimental): Participants are randomly assigned to receive either shockwave therapy or electromagnetic pulse therapy. Once assigned, the treatment method is fixed and continues for 12 weeks. From week 1 to week 12, participants receive either extracorporeal shockwave therapy or electromagnetic pulse therapy three times a week, totaling 36 sessions. After the completion of the 12-week treatment, the general rehabilitation program for lymphedema continues, conducted three times a week.
  Interventions: Device: Pulse electromagnetic field therapy

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — 2 times/week for 12 weeks
  Arms: ESWT therapy group
Device: Pulse electromagnetic field therapy — 2 times/week for 12 weeks
  Arms: PEMFT therapy group
Other: Rehabilitation — 2 times/week for 12 weeks
  Arms: General rehabilitation therapy

SUMMARY:
Lymphedema occurs not only in patients with breast cancer and gynecological cancers but also in those where lymphatic drainage is obstructed. Accumulation of lymphatic fluid within tissues results in limb swelling. Additionally, proteins present in lymphatic fluid might lead to fibrosis within tissues, causing various challenges for patients. The changes in volume and weight can significantly impact daily life activities such as eating, brushing teeth, and other routine tasks. Furthermore, it can lead to clothing difficulties and provoke unwanted attention due to aesthetic concerns.

Currently, there is no definitive treatment for lymphedema. However, prospective research has shown promising results in applying extracorporeal shock wave therapy (ESWT), originally used for musculoskeletal disorders like plantar fasciitis, tennis elbow, frozen shoulder, and non-union fractures, to lymphedema patients. Similarly, Pulse Electromagnetic Field Therapy (PEMFT), widely used for pain management and muscle strengthening, has the potential for treating lymphedema as it can enhance blood circulation and stimulate muscle contractions.

This research project aims to explore the effectiveness and sustainability of using ESWT and PEMFT for lymphedema patients. By applying these therapies to lymphedema patients, this study aims to evaluate their treatment outcomes and long-term effects.

DETAILED DESCRIPTION:
There is currently no cure for lymphedema. Literature review revealed extracorporeal shock wave therapy (previously applied to soft tissue diseases such as plantar fasciitis, tennis elbow, frozen shoulders, and poor fracture healing) showed positive therapeutic effect for patients with lymphedema.

Another widely used therapy for pain treatment and muscle strengthening is Pulse Electromagnetic Field Therapy (PEMFT), which has the potential to be used in the treatment of lymphedema due to its ability to increase blood circulation and stimulate muscle contractions.

This study design to evaluate the effect of extracorporeal shock wave therapy on patients with lymphedema, and further explore its therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 20 years old and have no significant cognitive, language comprehension, or communication issues, be able to understand and follow instructions, and sign the informed consent form.
* Individuals with lymphedema after treatment for breast cancer or gynecologic cancer are eligible (lymphedema is defined as a circumference difference of >2 cm in the same location on both limbs).
* You must be able to attend follow-up appointments at specific times during the 12 months of the trial, referred by a rehabilitation physician in the outpatient department.

Exclusion Criteria:

* The affected limb has unhealed open wounds, acute infections, or other conditions unsuitable for contact-based treatment.
* The affected limb has metastatic tumors.
* The affected limb has untreated deep vein thrombosis.
* Severe clotting abnormalities.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
circumference | every 1 week, through study completion, an average of 1 year
  Limb circumference
Thickness | every 1 week, through study completion, an average of 1 year
  thickness of skin and Subcutaneous tissue
Hardness | every 1 week, through study completion, an average of 1 year
  Hardness by shearwave elastography

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Yu Hoe, MD.,PhD., Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No